CLINICAL TRIAL: NCT04211675
Title: A Phase I/II Safety Lead in Study of Ex-Vivo Expanded Allogeneic Universal Donor TGFβi NK Cell Infusions in Combination With Irinotecan, Temozolomide, and Dinutuximab in Patients With Relapsed or Refractory Neuroblastoma: The Allo - STING Trial
Brief Title: NK Cells Infusions With Irinotecan, Temozolomide, and Dinutuximab
Acronym: STING
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000476
Record Dates: First submitted 2019-10-14; First posted 2019-12-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Relapsed Neuroblastoma; Refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — IL32 protein, human; Temozolomide; Irinotecan; dinutuximab; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): The planned therapy will involve 6 cycles of 21 days each consisting of irinotecan, temozolomide, dinutuximab, sargramostim, and natural killer (NK) cells.
  Treatment cycles will be repeated every 21 days based upon disease response and toxicity criteria. Tumor response will be assessed after Cycles 2, 4 and 6. Patients who do not experience dose-limiting toxicities and achieve complete response, partial response or stable disease may continue to receive the assigned therapy.
  Interventions: Biological: Natural Killer Cells; Drug: Temozolomide; Drug: Irinotecan; Drug: Dinutuximab; Drug: Sargramostim

INTERVENTIONS:
Biological: Natural Killer Cells — NK cells dose 1x 108 cells/ kg on day 8 of each cycle
Drug: Temozolomide — Temozolomide 100mg/m2/dose PO or IV daily on Days 1-5; if given orally, must be at least one hour prior to Irinotecan. For patients whose body surface area is <0.5m2, temozolomide dosing is based on body weight in (kg), at a dose of 3.3 mg/kg/dose.
  Other Names: Temodar
Drug: Irinotecan — Irinotecan 50mg/m2/dose IV daily on Days 1-5
  Other Names: Camptosar
Drug: Dinutuximab — Dinutuximab 17.5mg/m2/dose IV daily on Days 2-5
Drug: Sargramostim — Sargramostim 250mcg/m2/dose subcutaneous daily on Days 6-12
  Other Names: Leukine

SUMMARY:
This is a Phase 1 study with Phase 2 expansion cohort. Phase 1 will assess the safety and tolerability of universal donor TGFβi NK Cell in combination with irinotecan, temozolomide, and dinituximab. The phase 2 of the study will estimate the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Less than 30 years of age when registered on the study.
* Patients must have a histologic verification of neuroblastoma (NBL) or ganglioneuroblastoma or NBL cells in bone marrow with or without elevated urine catecholamines.
* Life expectancy >2 months, AND one of the following:

  * Recurrent disease; or
  * First episode of progressive disease (new lesion, increase in size, previous negative bone marrow) during initial multi-drug, induction myelosuppressive therapy; or
  * Primary resistant/refractory disease (partial, mixed, stable response criteria met) after completing at least 4 cycles of induction multi-drug induction chemotherapy
* One of the following:

  * Patients must have measurable or evaluable tumor defined as: a) Measurable tumor on MRI or CT obtained within 4 weeks prior to study entry; Measurable is defined as ≥ 10mm in at least one dimension AND that has positive uptake on I-123 MIBG scan ("MIBG avid") or demonstrates increased FDG uptake on 18F-FDG PET-CT or PET-MRI ("PET-avid"); OR b) Evaluable tumor by I-123 MIBG scan within 4 weeks prior to study entry, defined as positive uptake at a minimum of one site;
  * Measurable or evaluable disease must represent recurrent disease after therapy completion or progressive disease on therapy or refractory disease during induction;
  * Patients with refractory disease that are not avid on MIBG scan and do not have increased FDG uptake on PET must have biopsy proven viable NBL;
  * New soft tissue sites that are MIBG avid or PET avid do not require biopsy as long as initial histologically-confirmed NBL diagnosis prior to current therapy
* Patients must have progressed during or following completion of frontline therapy. Agents considered to be a part of frontline therapy would include chemotherapy, radiation therapy, autologous stem cell transplantation, retinoids, immunotherapy with anti GD2 agents, cellular therapies, or I-131 MIBG, and frontline therapy is defined as any combination of these agents defined in published regimens or current cooperative group clinical trials for the successful treatment of that cancer. Therapy may not have been received more recently than the timeframes defined below:

  * Myelosuppressive chemotherapy: At least 14 days since completion of myelosuppressive therapy
  * Biologic: At least 7 days since completion of therapy with non-myelosuppressive biologic or retinoid
  * Radiation: At least 4 weeks since completion of radiation to any site identified as a target lesion. Palliative radiation is allowed to sites not used to measure response
  * Stem Cell Transplant (SCT): At least 6 weeks after autologous stem cell transplant or stem cell infusions as long as hematologic criteria have been met
  * 131I-MIBG Therapy: At least 6 weeks after therapeutic MIBG treatment
  * Cellular therapies: At least 6 weeks after any cellular therapy treatment (e.g., prior NK, CAR-T therapy)

Subjects who have previously received anti-GD2 monoclonal antibodies for biologic therapy or for tumor imaging are eligible.

Subjects who have received autologous marrow infusions or autologous stem cell infusions that were purged using monoclonal antibody linked to beads are eligible.

No treatment with irinotecan and/ or temozolomide within the last 6 months.

* Adequate bone marrow function, defined as:

  * Peripheral absolute neutrophil count (ANC) ≥500/microL. Patients must not have received long-acting myeloid growth factors (e.g., Neulasta) within 14 days or short-acting myeloid growth factors (e.g., Neupogen) within 7 days of study entry.
  * Platelet count ≥50,000/microL (transfusion independent for at least 1 week)
* Adequate renal function defined as:

  * Creatinine clearance or estimated radioisotope GFR ≥70 ml/min/1.73m2 or
  * Serum creatinine < 2x upper limit of normal (ULN) based on age/gender
* Adequate liver function defined as:

  * Total bilirubin <1.5x ULN for age AND
  * SGPT (ALT) ≤5x ULN for age (or ≤225 U/L). For purpose of this study, the ULN for SGPT (ALT) is 45 U/L.
* Adequate central nervous system function defined as:

  * Patients with seizure disorders may be enrolled if seizures are well controlled on anti-convulsants
  * CNS toxicity ≤ Grade 2
* Adequate cardiac function defined as:

  * Shortening fraction of ≥ 27% by ECHO OR
  * Ejection fraction ≥ 50% by ECHO or gated radionuclide study
* Adequate pulmonary function defined as:

  * No evidence of dyspnea at rest, no exercise intolerance, no chronic oxygen requirement, and room air pulse oximetry > 94% if there is a clinical indication for pulse oximetry

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients with elevated catecholamines (>2x ULN) only.
* Patients must not have received 0.5 mg/ kg/ day (prednisone equivalent) doses of systemic steroids for at least 7 days prior to enrollment.
* Patients must not have received CYP3A4 inducer or inhibitor for at least 7 days prior to study enrollment.
* Patients must not have been diagnosed with any other malignancy.
* Patients must not have > Grade 2 diarrhea.
* Patients must not have uncontrolled infection.
* Patients with history of Grade 4 allergic reactions to anti-GD2 antibodies or reactions that required discontinuation of anti-GD2 therapy.
* Patients with a significant illness that is not covered by the exclusion criteria or that is expected to interfere with the action of study agents or to increase the severity of the toxicities experienced from the study treatment.

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
NK cells safety and tolerability: Number of participants with treatment-related adverse events and toxicities | 12 months
  Number of participants with treatment-related adverse events and toxicities as assessed by CTCAE v4.0
Response to NK Cell treatment as determine by CT/MRI imaging | 24 months
  To estimate the response to treatment, as determined by disease status evaluated using CT/MRI scans through the measuring tool RECIST.
Response to NK Cell treatment as determine by MIBG scans imaging | 24 months
  To estimate the response to treatment, as determined by disease status evaluated using MIBG scans through the Curie score system.
Response to NK Cell treatment as determine by bone marrow aspiration | 24 months
  To estimate the response to treatment, as determined by disease status evaluated using bone marrow aspiration and biopsy through H&E stain. RECIST.

SECONDARY OUTCOMES:
Toxicity Definition of NK cells | 36 months
  Toxicity will be graded using the CTCAE criteria, version 5.0. All grade 3+ toxicities will be reviewed for attribution.

OTHER OUTCOMES:
Assessment of the phenotype of expanded NK cells for neuroblastoma patients | 36 months
  NK cell phenotypes will be measured by mass cytometry (unit of measure= % of nucleated cells)
Assessment of function of expanded NK cells for neuroblastoma patients | 36 months
  NK cell functional potency will be measured as cytotoxicity by calcien- AM cytotoxicity assays (unit of measure= % of patietns with complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD), or progressive disease (PD) with calculated 95% confidence intervals)
In vivo persistence of NK cells after adoptive transfer. | 36 months
  To assess in vivo persistence of expanded NK cells after adoptive transfer by assessing NK cell number and phenotype in peripheral blood using mass cytometry.
Correlation of persistence of NK cells after adoptive transfer with clinical outcomes | 36 months
  Clinical outcomes will be assessed by disease response using CT/MRI scans, I-123 metaiodobenzylguanidine (MIBG) scans, and bone marrow aspiration and biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ranalli, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States